CLINICAL TRIAL: NCT04273724
Title: A Pilot Study of Early Intervention for Impairments Identified During Comprehensive Geriatric Assessment in Patients With Muscle-invasive Bladder Cancer
Brief Title: Early Intervention for Impairments Identified During Comprehensive Geriatric Assessment in Patients With Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left and research was discontinued.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 1946
Record Dates: First submitted 2020-02-05; First posted 2020-02-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Geriatric oncology; Comprehensive geriatric assessment; Patient-reported outcomes; Muscle-invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geriatric assessment guided interventions (Experimental)
  Interventions: Other: Targeted Interventions for Impairments Identified During Geriatric Assessment

INTERVENTIONS:
Other: Targeted Interventions for Impairments Identified During Geriatric Assessment — Participants will be referred for specific evidence-based interventions based on impairments identified during a baseline comprehensive geriatric assessment.

SUMMARY:
A Comprehensive Geriatric Assessment (CGA) is a set of tests used to evaluate a patient's medical, social, and functional status, and can identify impairments in these domains that may not be noticed otherwise. Prior studies have shown that a CGA can accurately predict which patients are more likely to have serious side effects from cancer treatment. However, it is unknown whether interventions can be done to address the impairments found during a CGA in order to reduce the risk of these side effects. This pilot study will test the feasibility of targeted interventions for deficits identified during a CGA in patients 65 years or older with bladder cancer that have not yet started treatment.

DETAILED DESCRIPTION:
This study will enroll patients with muscle-invasive bladder cancer that have not yet started systemic cancer treatment. The participants will complete a CGA and patient-reported outcome (PRO) measures at baseline. Based on any impairments found during the CGA, participants will be referred to specialists to help address these difficulties. Participants will complete the CGA and PRO measures again at 3 months and 1 year after the initial assessment. The goal of this study is to see if patients with advanced bladder cancer are interested in referrals to specialists to address their impairments, and whether participants attend those appointments.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Confirmed diagnosis of muscle-invasive bladder cancer
* Plan to undergo systemic treatment but have not yet started therapy

Exclusion Criteria:

* Must be able to read English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Patient interest in impairment-directed interventions | 1 year
  To establish patient interest in referral for interventions based on impairments found during geriatric assessment within an outpatient genitourinary oncology clinic. Success will be at least 75% of patients accepting referral for indicated interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No